CLINICAL TRIAL: NCT01549977
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Assess the Effect of Febuxostat 80 mg Once Daily Compared to Placebo on Exercise Tolerance in Subjects With Chronic Stable Angina
Brief Title: Effect of Febuxostat Compared to Placebo on Exercise Tolerance in Participants With Chronic Stable Angina
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision (please see below)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_207; U1111-1125-1278 (Registry Identifier: WHO)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-10

CONDITIONS: Angina
Keywords: Drug Therapy
MeSH Terms: conditions — Angina Pectoris | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat 80 mg (Experimental): Febuxostat 80 mg, tablets, orally, once daily for up to 12 weeks.
  Interventions: Drug: Febuxostat
- Placebo (Placebo Comparator): Febuxostat placebo-matching tablets, orally, once daily for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat tablets
  Other Names: TMX-67; Uloric
  Arms: Febuxostat 80 mg
Drug: Placebo — Febuxostat placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of febuxostat, once daily (QD), compared to placebo as an add on to stable anti-anginal therapy, on the total exercise time of participants with Chronic Stable Angina.

DETAILED DESCRIPTION:
This is a phase 2 multicenter, randomized, placebo-controlled double-blind study. This study is comprised of a single-blind placebo run-in qualifying phase lasting approximately 3 weeks and a double-blind treatment phase lasting 12 weeks. A safety follow-up visit is scheduled for 2 weeks after last dose of study drug.

All participants will undergo 3 visits during a 3 week, run-in phase (Days -21 to Day 1). During the run-in phase, all participants will receive single-blind placebo. Two exercise treadmill tests (ETTs) will be conducted using the modified Bruce Protocol at Day -14 and at Day -7. The results from the Day -7 ETT will be considered as Baseline.

A total of approximately 100 participants will be randomized 1:1 to receive either febuxostat 80 mg once daily (QD) or placebo QD in a double-blind treatment for 12 weeks, and 5 more visits.

All participants will complete the Seattle Angina Questionnaire (SAQ) and Euroqol 5 dimension (EQ-5D) quality-of-life measurements at Day 1, Week 6 and Week 12/Early Termination (ET) Visit. The investigator will also rate the overall severity of the participant's angina at each visit based on the Canadian Cardiovascular Society Grading of Angina (CCSGA).

This 12-week phase 2 proof-of-concept study was designed to assess the effect of febuxostat as an add-on to stable anti-anginal therapy on the total exercise time of participants with chronic stable angina and a serum urate ≥5 mg/dL. At this time, Takeda has decided to terminate the study for business reasons.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative, signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant has an serum urate (sUA) ≥5.0 mg/dL.
4. The participant has a history of angina, defined as:

   1. Minimum of 3-month history of stable angina (at least 2 episodes of chest pain or anginal equivalent in the past 30 days); AND
   2. Receiving at least one chronic anti-ischemic medication(s), including beta blockers, calcium channel blockers and long acting nitrates (doses must be stable for at least 30 days prior to Screening [Day -21]); AND
   3. Coronary artery disease, as defined by:

      * ≥50 % stenosis of ≥1 major coronary artery confirmed by angiography; OR
      * Documented prior myocardial infarction (MI) by enzymes/electrocardiogram (ECG) changes; OR
      * Documented myocardial imaging stress test; OR
      * Prior history of coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) greater than 3 months prior to Screening Day -21.
5. The participant has estimated glomerular filtration rate (eGFR) >30 mL/min by Modification of Diet in Renal Disease (MDRD) at the Screening visit Day -21.
6. The participant has a normal/controlled blood pressure at Day 1/Randomization, as defined by the mean of three sitting blood pressures not exceeding 140/90.
7. The participant is male or female and aged 18 to 85 years, inclusive.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
9. Participant is on stable (30 days) medication doses prescribed for any underlying medical condition (ie; hypertension, angina) and will remain on stable doses throughout the study duration.
10. Participant is able to take, in an ongoing manner, nitroglycerine for anginal symptoms.
11. Symptom-limited exercise duration, during ETT at Day -14 and Day -7, on the modified Bruce Protocol.
12. Exercise duration for the two ETTs at Day -14 and Day -7 did not differ by more than 20% of the longer of the two times, and did not differ by more than 60 seconds. To be confirmed by the Core ECG Lab prior to the subject being randomized.
13. Definite ECG signs of ischemia during the ETT at both Day -14 and Day -7 (i.e., 1 additional mm of horizontal or down-sloping ST-segment depression beyond baseline and ≥1 mm below the isoelectric line) are present in at least one standard ECG lead during ETT. The Day -7 ≥1 mm ST-segment depression must be verified by the Core ECG Lab prior to participant being randomized.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to Screening Day -21.
2. The participant has received allopurinol or febuxostat in a previous clinical study or as a therapeutic agent.
3. The participant has gout or secondary hyperuricemia (e.g., due to myeloproliferative disorder, or organ transplant) or has experienced a gout flare.
4. The participant has a history of xanthinuria.
5. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
6. The participant has a history of hypersensitivity or allergies to febuxostat or nitroglycerine.
7. The participant has hemoglobin <10 g/L at Screening Day -21.
8. The participant has a systolic blood pressure of less than 100 mmHg.
9. The participant has a blood pressure of greater than 200/100 at any Screening or Run-in visit.
10. The participant has a history or clinical manifestations of a significant medical condition that might affect his/her ability to complete the study.
11. The participant has any of the following at any Screening or Run-in visit:

    1. Resting ST-segment depression ≥1 mm in any lead.
    2. Left bundle-branch block.
    3. New York Heart Association Class III or IV heart failure.
    4. Acute coronary syndrome or a coronary revascularization procedure within 3 months of Screening.
    5. Wolff-Parkinson-White syndrome.
    6. Pacemaker or implantable cardioverter defibrillator.
    7. Arrhythmias (i.e., SVT, atrial fibrillation/flutter, VT, or rate related bundle branch blocks).
    8. Left ventricular hypertrophy with repolarization abnormalities.
12. The participant has a recent history (within the last 3 months) of myocardial infarction, heart failure, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
13. The participant has a contraindication for using nitrates (severe anemia, increased intracranial pressure, and those with a known sensitivity or hypersensitivity to nitroglycerin or its ingredients, or other nitrates or nitrites; concomitant use either regularly and/or intermittently, with phosphodiesterase type 5 (PDE5) inhibitors).
14. The participant has unstable angina that:

    1. Occurs when the participant is at rest.
    2. Is prolonged, usually greater than 20 minutes.
    3. Occurs with increasing in intensity, duration, and/or frequency.
    4. Responds poorly to nitroglycerin (i.e., does not go away after three doses of nitroglycerin or returns after the nitroglycerin helped at first).
15. The participant is unable to exercise sufficiently to complete ETT due to leg claudication, arthritis, deconditioning, or associated pulmonary disease.
16. The participant has severe or critical valvular disease documented by echocardiogram, or congenital heart disease.
17. The participant has left ventricular ejection fraction (LVEF) less than 35%, as documented by echocardiogram or angiography.
18. The participant has clinically significant cardiac conduction defects (i.e., second- or third-degree atrioventricular block, sick sinus syndrome or a QTc >500 msec) at Day -21.
19. The participant has active acute myocarditis/pericarditis within the 3 months prior to Screening Day -21.
20. The participant has hypertrophic cardiomyopathy.
21. The participant has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level of greater than 2.0 times the upper limit of normal, has active liver disease, or jaundice.
22. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the Screening Visit.
23. The participant is required or expected to require excluded medications digoxin and digoxin-containing compounds.
24. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
25. The participant has participated in another clinical study within the past 30 days.
26. The participant has a history of extracorporeal external counterpulsation treatment for chronic stable angina within 3 months prior to screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (21):
- United States (21):
  - Carmichael, California
  - Fresno, California
  - Irvine, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Tampa, Florida
  - Dunwoody, Georgia
  - Suwanee, Georgia
  - Lexington, Kentucky
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - Salisbury, North Carolina
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Tipton, Pennsylvania
  - San Antonio, Texas
  - Manassas, Virginia
  - Port Orchard, Washington
  - Madison, Wisconsin

REFERENCES:
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with a diagnosis of chronic stable angina were enrolled in 1 of 2 treatment groups, placebo or febuxostat 80 mg once daily.
Period: Overall Study
Arm/Group | Febuxostat 80 mg | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 80 mg | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: participants]
  18 to 65 years | 0 |  | 0
  ≥ 65 years | 1 |  | 1
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Exercise Treadmill Testing (ETT) Duration at Week 12
Description: The change between the duration of ETT at Week 12 relative to Baseline. ETTs were conducted using the modified Bruce Protocol. Participants exercised on a treadmill, starting at 1.7 mph and 0% incline. The intensity of exercise (speed and/or incline) was increased at 3 minute intervals.
Time Frame: Baseline and Week 12
Population: This analysis was not performed since only one participant completed the study prior to study termination.
Arm/Group | Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Time to Onset of Angina During ETT at Week 12
Description: The change between the time to onset of angina during the exercise treadmill test (ETT) at Week 12 relative to Baseline.
Time Frame: Baseline and Week 12
Population: This analysis was not performed since only one participant completed the study prior to study termination.
Arm/Group | Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Time to Onset of ≥1 mm ST-segment Depression During ETT at Week 12
Description: The change between the time to onset of ≥1 mm ST-segment depression during exercise treadmill test (ETT) at Week 12 relative to Baseline. ST-segment is measured by electrocardiography (ECG) and represents the interval between ventricular depolarization and repolarization.
Time Frame: Baseline and Week 12
Population: This analysis was not performed since only one participant completed the study prior to study termination.
Arm/Group | Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Maximum ST-segment Depression During ETT at Week 12
Description: The change between the maximum ST-segment depression during ETT at Week 12 relative to Baseline. ST-segment is measured by electrocardiography (ECG) and represents the interval between ventricular depolarization and repolarization.
Time Frame: Baseline and Week 12
Population: This analysis was not performed since only one participant completed the study prior to study termination.
Arm/Group | Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Stopping ETT Due to Angina at Week 12
Description: The percentage of participants who had to stop exercise treatment testing (ETT) due to experiencing angina symptoms at Week 12.
Time Frame: Week 12
Population: This analysis was not performed since only one participant completed the study prior to study termination.
Arm/Group | Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Febuxostat 80 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg (N=1) | Placebo (N=0)
Blood creatinine increased (Investigations) | 1 | 0
Urinary sediment present (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Insufficient data to publish.